CLINICAL TRIAL: NCT01521611
Title: Radiolabelled Anti-CD66 Monoclonal Antibody in the Conditioning Regimen Prior to Haematopoietic Stem Cell Transplantation: Phase I Study in Patients With Poor-risk Disease.
Brief Title: Targeted Radiotherapy in HSCT for Poor Risk Haematological Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Royal Free and University College Medical School (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN0227
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Acute Leukaemia; Chronic Leukaemia; Myeloma; Lymphoma
Keywords: Radioimmunotherapy; Transplant; Bone Marrow Transplant (BMT); yttrium; indium
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targeted radiotherapy (Experimental): Patients receive therapy with an yttrium-90 labelled anti-CD66 following favourable dosimetry with the same antibody radiolabelled with indium-111.
  Interventions: Radiation: Targeted radiotherapy

INTERVENTIONS:
Radiation: Targeted radiotherapy — Yttrium-90 labelled anti-CD66 monoclonal antibody.
  Other Names: Y-90-anti-CD66

SUMMARY:
To determine whether a radiolabelled antibody that targets the bone marrow (the 'anti-CD66') can be administered safely to patients as part of the preparative treatment prior to haematopoietic stem cell transplantation ('a bone marrow transplant'). Can the radiolabelled antibody be shown to effectively target the bone marrow in these patients. If it can, could this result in better outcomes after transplantation.

DETAILED DESCRIPTION:
The aim of this clinical research study is to establish whether a radiolabelled antibody can be used to safely deliver radiotherapy to the bone marrow prior to stem cell transplantation for haematological malignancies.

With current chemotherapy regimens 60-90% of adult patients with acute leukaemia (AML and ALL) achieve a complete remission. However in a significant proportion of these patients the disease will recur. Although allogeneic and autologous bone marrow or peripheral blood haematopoietic stem cell transplantation (HSCT) are established as effective treatment options for haematological malignancies, resulting in long term disease free survival in a significant proportion of patients, the results of transplantation for patients with poor risk disease are disappointing. Further intensification of the treatment used prior to transplantation has been shown to reduce the risk of relapse, but the toxicity of the drugs or external beam radiotherapy causes an increase in transplant related deaths. The introduction of reduced intensity conditioning protocols allows the use of HSCT for older patients or those with significant additional medical problems but retrospective analysis indicates an increased rate of relapse. This is the 'Transplantation dilemma' - how to reduce the risk of disease relapse by intensifying therapy, but without an increase in toxicity to other organs causing an increase in transplant related deaths in remission.

Normal haematopoietic tissue and the malignant cells arising from it are very radiosensitive. Theoretically intensification of the conditioning therapy, particularly total body irradiation (TBI), prior to transplantation could increase tumour reduction leading to improved disease free survival rates for patients with poor risk disease. Targeted radiotherapy could allow treatment intensification without the toxicity to non-haematological tissues. In addition, the continuous, low dose rate delivered by the natural decay of a targeted radionuclide may have a greater destructive effect upon tumour cells than single dose or fractionated external beam radiation.

ELIGIBILITY:
Inclusion Criteria:

1. An underlying haematological malignancy including acute myeloid leukaemia in first complete remission (CR1) but with poor prognostic features or in >CR1 or in relapse; acute lymphoblastic leukaemia; transformed myelodysplasia, chronic myeloid leukaemia (accelerated phase or blast transformation, poor response or intolerance of tyrosine kinase inhibitors), myeloma. Patients may be in remission, partial remission or relapse.
2. No concurrent or recent (within 3 weeks) chemotherapy for the underlying haematological condition
3. For patients with relapsed leukaemia, bone marrow (BM) blasts must represent < 20% of BM nucleated cells.
4. Although the BM remission status is not important, patients must have cellularity > 10%.
5. As malignant plasma cells may or may not express CD66 antigens, patients with myeloma must have less than 30% plasma cells (as a percentage of total nucleated cells) in the BM at the time of the study.
6. Age = or >18 yrs.
7. WHO performance status of 0, 1 or 2 (Appendix 5).
8. Predicted life-expectancy of greater than four months.
9. Patients must be negative for human anti-mouse antibodies (HAMA).
10. Peripheral blood counts:

    Wbc < 30 x 10e9/l (absolute neutrophil count >0.5 x 10e9/L) platelets > 50 x 10e9/l (platelet support is permitted)
11. Biochemical indices:

    Plasma creatinine < 120 micromol/l (or creatinine clearance or Ethylene diamine tetra acetic acid (EDTA) clearance > 50 ml/min) Plasma bilirubin < 30 micromol/l Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) no more than 2.5 x upper limit of the normal range.
12. Patient must be able to provide written informed consent.

Exclusion Criteria:

1. Any serious intercurrent disease.
2. Patients with BM cellularity < 10%.
3. History of atopic asthma, eczema or allergy to rodent protein, confirmed history of severe allergic reactions to penicillin or streptomycin.
4. Positive Human anti-murine antibodies (HAMA).
5. Patients unable to provide informed consent or who are unable to co-operate for reasons of poor mental or physical health.
6. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Toxicities related to radiolabelled antibody. | Up to 1 year post transplant World Health Organisation (WHO) toxicity criteria
  To determine the maximum tolerated dose (MTD) of targeted radiotherapy delivered by a murine anti-CD66 monoclonal antibody radiolabelled with yttrium-90 (Y-90) and determine the dose-limiting toxicity (DLT) in patients with haematological malignancies who are undergoing haematopoietic stem cell transplantation.
  Toxicities are assessed using WHO Toxicity Scale with 28 parameters.

SECONDARY OUTCOMES:
Dosimetry model | 5 days post infusion of an Indium-111 radiolabelled anti-CD66
  Dosimetry is determined by whole body and SPECT-CT of the thorax and abdomen on days 1, 2, 4 and 5 post infusion of an indium-111 radiolabelled anti-CD66. Dosimetry determines whether patients proceed to therapy with the yttrium-90 labelled anti-CD66.

CONTACTS AND LOCATIONS:
Overall Officials: Kim H Orchard, MBBS PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Southampton University Hospitals NHS Trust, Southampton, Hampshire
  - Royal Free Hospital and University College London, London

IPD SHARING:
Plan to Share IPD: No
Trial fully recruited. Data will be summarised upon completion of study.

REFERENCES:
- [Derived] Orchard K, Langford J, Guy M, Lewis G, Michopoulou S, Cooper M, Zvavamwe C, Richardson D, Lewington V. Efficient bone marrow irradiation and low uptake by non-haematological organs with an yttrium-90-anti-CD66 antibody prior to haematopoietic stem cell transplantation. Bone Marrow Transplant. 2024 Sep;59(9):1247-1257. doi: 10.1038/s41409-024-02317-z. Epub 2024 Jun 12. PMID 38867006